CLINICAL TRIAL: NCT00744055
Title: The Use of Prazosin for Treatment of Patients With Alcohol Dependence (AD) and Post Traumatic Stress Disorder (PTSD).
Brief Title: Prazosin for Treatment of Patients With Alcohol Dependence (AD) and Post Traumatic Stress Disorder (PTSD).
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0801003450
Record Dates: First submitted 2008-08-28; First posted 2008-08-29 (Estimated); Results first posted 2016-01-18 (Estimated); Last update posted 2020-03-19 (Actual); Status verified 2020-03

CONDITIONS: Alcohol Dependence; Stress Disorders, Post-Traumatic
Keywords: alcohol dependence; post traumatic stress disorder; treatment; prazosin
MeSH Terms: conditions — Alcoholism; Stress Disorders, Post-Traumatic | interventions — Prazosin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Prazosin (Experimental): prazosin (16mg/day)
  Interventions: Drug: Prazosin
- Placebo (Placebo Comparator): Placebo in identical looking capsule blister packs
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Prazosin — prazosin (16mg/day) 2 times a day
  Other Names: Minipress
  Arms: Prazosin
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
Prazosin is an alpha-1 adrenergic receptor antagonist that has been used successfully in the treatment of trauma nightmares and sleep disturbance in combat veterans with PTSD, and alcohol dependence.

The objective of this study is to evaluate the efficacy of prazosin (16mg) versus placebo in reducing alcohol consumption and decreasing symptoms of PTSD in patients with comorbid AD and PTSD.

DETAILED DESCRIPTION:
Background:

There is a high rate of comorbidity with alcohol dependence (AD) and post traumatic stress disorder (PTSD). The rates of PTSD among individuals with AD are at least twice as high as those in the general population. In addition, alcohol dependence is the most common comorbid condition in men with PTSD. Despite this, little is known about how to best treat individuals with comorbid AD and PTSD. The use of an alpha-1 adrenergic receptor antagonist represents a novel approach to treatment that may target symptoms of both AD and PTSD. There is evidence of common neurobiological mechanisms that underlie both AD and PTSD. Prazosin is an alpha-1 adrenergic receptor antagonist that has been used successfully in the treatment of trauma nightmares and sleep disturbance in combat veterans with PTSD, and alcohol dependence.

Objective:

The objective of this study is to evaluate the efficacy of prazosin (16mg) versus placebo in reducing alcohol consumption and decreasing symptoms of PTSD in patients with comorbid AD and PTSD. Methods: Thirty participants with a current diagnosis of AD and PTSD will be enrolled in a 13-week trial. They will be assigned, in a double-blind fashion, to either prazosin or placebo. Significance: This project will be the first to compare prazosin to placebo as effective treatments for reducing alcohol consumption and PTSD symptoms in patients with both AD and PTSD.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females between the ages of 21-65 years old.
2. Current alcohol dependence, as determined by a structured clinical interview (Structured Clinical Interview for DSM-IV Axis I Disorders) (SCID) (First et al. 1996).
3. Current PTSD as determined by the Clinician Administered PTSD Scale for DSM-IV(CAPS) (Blake et al. 1995).
4. Patients with current alcohol dependence, with at least one recent episode of heavy drinking (defined as 5 or more drinks per drinking episode) over the past 14 days.
5. Medically and neurologically healthy on the basis of history, physical examination, EKG, screening laboratories (CBC w/ differential, TSH, Free-T4, ASAT, ALAT, GGT, BUN, creatinine, calcium, phosphorous, magnesium, total protein, albumin, electrolytes, VDRL, urinalysis, beta-HCG).
6. For women, negative pregnancy test and use of acceptable method of contraception.

Exclusion Criteria:

1. Females who are pregnant or lactating.
2. Individuals with a current unstable medical condition such as neurological, cardiovascular, endocrine, renal, liver, or thyroid pathology (LFT 5 times normal, abnormal BUN and creatinine, and unmanaged hypertension with BP more than 200/120) which in the opinion of the physician would preclude the patient from fully cooperating or be of potential harm during the course of the study.
3. Patients who meet current SCID criteria for the following major Axis I diagnoses (Bipolar Disorders, Schizophrenia and Schizophrenia-type Disorders).
4. History of substance dependence (other than alcohol, cocaine, tobacco or cannabis) by DSM-IV criteria in the last 30 days.
5. Individuals taking mood stabilizers and antipsychotic medications.
6. Individuals with a history of sensitivity to quinazolines or prazosin.
7. Individuals taking medications thought to influence alcohol consumption (naltrexone, disulfiram, acamprosate).
8. Individuals taking adrenergic medication (e.g. clonidine).
9. Agents that may interact with prazosin such as drugs with CNS depressant effects including tizanidine and xyrem.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2009-01; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ismene Petrakis, MD, Principal Investigator — Yale University
Locations (1):
- VA Connecticut Healthcare System, West Haven, Connecticut, United States

REFERENCES:
- [Derived] Gandelman E, Petrakis I, Kachadourian L, Ralevski E. Negative Affect Intensity and Hostility in Individuals With Alcohol Use Disorder With or Without Posttraumatic Stress Disorder. J Dual Diagn. 2018 Apr-Jun;14(2):96-101. doi: 10.1080/15504263.2018.1434264. Epub 2018 Apr 25. PMID 29461925

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Randomization was conducted by the pharmacy using a 1:1 randomization in blocks of 4 and stratified by site, gender.
  Completers were defined as subjects for whom we had complete data at the end of the treatment period (week 12) whether they remained on medication or not.
Period: Overall Study
Arm/Group | Prazosin | Placebo
Started | 50 | 46
Completed | 43 | 32
Not Completed | 7 | 14
Not completed — Withdrawal by Subject | 6 | 9
Not completed — Lack of Efficacy | 0 | 1
Not completed — Physician Decision | 0 | 2
Not completed — Protocol Violation | 1 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Population: Veterans
Groups:
- Prazosin; Placebo: men or women, ages of 21-65, met DSM-IV criteria for current PTSD and alcohol dependence (AD) (determined by structured clinical interview)
- Total: Total of all reporting groups
Arm/Group | Prazosin | Placebo | Total
Number analyzed (Participants) | 50 | 46 | 96
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.5 (13.2) | 43.40 (12.95) | 43.96 (12.96)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 | 6
  Male | 46 | 44 | 90
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 40 | 38 | 78
  Non-Caucasian | 10 | 8 | 18
PTSD Symptoms [Mean (Standard Deviation); unit: units on a scale] — Clinician-Administered PTSD Scale for DSM-IV (CAPS-IV). The scale consists of 30 questions on a scale from 0-4.
  The lowest possible score is 0 and the highest possible score is 120. A higher score is associated with higher severity of PTSD. The score is interpreted as follows: 0-19=Asymptomatic/few symptoms 20-39=Sub-threshold/mild PTSD 40-59=Threshold PTSD/moderate 60-79=Severe PTSD >80=Extreme PTSD
  units on a scale | 71.86 (20.32) | 75.86 (14.44) | 73.7 (17.86)
Average Drinks Per Drinking Day [Mean (Standard Deviation); unit: drinks per day] | 17.33 (10.73) | 21.90 (13.24) | 19.53 (8.21)

OUTCOME MEASURES:

1. Primary Outcome: Number of Drinking Days
Description: Using the Timeline Follow Back method, a calendar method for assessing drug and alcohol use
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Prazosin | Placebo
Number analyzed (Participants) | 50 | 46
days | 11.04 (18.86) | 9.21 (16.64)

2. Primary Outcome: Clinician-Administered PTSD Scale
Description: Clinician-Administered PTSD Scale for DSM-5 (CAPS-5). A higher score is associated with higher severity of PTSD. The score is interpreted as follows: 0-19=Asymptomatic/few symptoms 20-39=Sub-threshold/mild PTSD 40-59=Threshold PTSD/moderate 60-79=Severe PTSD >80=Extreme PTSD
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Prazosin | Placebo
Number analyzed (Participants) | 50 | 46
units on a scale | 37.94 (37.62) | 37.93 (41.13)

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Prazosin | Placebo
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/46
Other Adverse Events (participants affected / at risk) | 11/50 | 8/46
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Prazosin (N=50) | Placebo (N=46)
Alcohol Relapse (Psychiatric disorders) | 5 | 7
Homocidal Ideation (Psychiatric disorders) | 0 | 1
Partial thrombus (Vascular disorders) | 1 | 0
Chest Pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Appendicitis (Gastrointestinal disorders) | 1 | 0
Fainting (General disorders) | 1 | 0
Falling (General disorders) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes